CLINICAL TRIAL: NCT05799170
Title: Evaluation of the Effectiveness of a Regional Trauma Care System for the Treatment of Patients With Severe Trauma: Protocol for a Prospective, Multicenter, Stepped-wedge Cluster-randomized Controlled Clinical Trial
Brief Title: Evaluation of the Effectiveness of a Regional Trauma Care System for the Treatment of Patients With Severe Trauma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Feifei Jin, Research assistant, Peking University People's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RT study
Record Dates: First submitted 2023-03-09; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Study intervention is the establishment of in-hospital trauma treatment centers and the formation of regional trauma care system. Regional trauma care system refers to both the establishment of unified and standardized pre-hospital and in-hospital trauma triage and injury classification warning mechanism and the development of unified trauma treatment process and standard in a main government district (population within 1 million), with secondary general hospitals and above that have strong treatment capability as the trauma treatment centers. Regional trauma care system will strengthen both pre-hospital emergency care and in-hospital emergency treatment while reinforcing the information exchange between in-hospital emergency treatment and specialized treatment.
  Interventions: Other: regional trauma care
- usual care (No Intervention): usual care/standard of care no intervention implemented

INTERVENTIONS:
Other: regional trauma care — Study intervention is the establishment of in-hospital trauma treatment centers and the formation of regional trauma care system. Regional trauma care system refers to both the establishment of unified and standardized pre-hospital and in-hospital trauma triage and injury classification warning mechanism and the development of unified trauma treatment process and standard in a main government district (population within 1 million), with secondary general hospitals and above that have strong treatment capability as the trauma treatment centers. Regional trauma care system will strengthen both pre-hospital emergency care and in-hospital emergency treatment while reinforcing the information exchange between in-hospital emergency treatment and specialized treatment. Taking 5 to 6 hospitals with certain trauma treatment capacity as the trauma treatment point, the trauma treatment network is formed relying on the treatment point hospitals within the range of one trauma treatment center.
  Arms: intervention

SUMMARY:
Severe trauma imposes a heavy burden to society and family because of its high mortality and disability rate. Based on the implementation plan of "one region", "two links", and "three teams", the Trauma Medicine Center of Peking University People's Hospital has constructed regional trauma care system that is suitable for China's national conditions. The primary objective of this trial is to evaluate the effectiveness of the regional trauma care system on the treatment of patients with severe trauma in China.This study is a prospective, multicenter, stepped-wedge cluster-randomized controlled clinical trial.

DETAILED DESCRIPTION:
Background: Severe trauma imposes a heavy burden to society and family because of its high mortality and disability rate. Based on the implementation plan of "one region", "two links", and "three teams", the Trauma Medicine Center of Peking University People's Hospital has constructed regional trauma care system that is suitable for China's national conditions. The primary objective of this trial is to evaluate the effectiveness of the regional trauma care system on the treatment of patients with severe trauma in China.

Methods: This study is a prospective, multicenter, stepped-wedge cluster-randomized controlled clinical trial. Twenty hospitals are selected based on specific eligibility criteria. After the baseline period, 5 randomization steps with 4 hospitals per step will be conducted. Each hospital will gradually enter intervention period in the randomized order for the implementation of regional trauma care system. The initial 1-month is considered as the intervention transition period, during which hospitals are modified and healthcare workers are trained according to the requirements of the regional trauma care system.

Conclusion: This is the first study assessing the effectiveness of the regional trauma care system on the treatment of patients with severe trauma with the conduction a prospective study in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-60 years old, with no restriction on gender;
2. Severe trauma, including trauma patients with ISS score ≥ 16;
3. Time from trauma to admission <24h.

Exclusion Criteria:

1. Patients who complicated with underlying diseases, such as malignant tumor and diabetes mellitus;
2. Patients with important organ dysfunction before trauma;
3. The investigator considers not appropriate for enrollment. -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3200 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the mortality of patients with severe trauma | one week
  The primary efficacy indicator is the mortality of patients with severe trauma at one week after trauma treatment. Mortality is defined as the percentage of patients with severe trauma who die after trauma treatment to the total number of patients with severe trauma receiving treatment.

IPD SHARING:
Plan to Share IPD: No